CLINICAL TRIAL: NCT00005986
Title: Autologous Transplantation for Chronic Myelogenous Leukemia Using Retrovirally Marked Peripheral Blood Progenitor Cells Obtained After In Vivo Cyclophosphamide/G-CSF Priming
Brief Title: Chemotherapy, Filgrastim and Peripheral Stem Cell Transplantation in Patients With Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator left the university.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Catherine Verfaillie, MD
Purpose: Treatment
Other Study IDs: CDR0000067974; UMN-MT-9507 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2000-07-05; First posted 2004-02-12 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Busulfan; Cyclophosphamide; Filgrastim; Interferon-alpha; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: filgrastim
Drug: recombinant interferon alfa
Procedure: in vitro-treated peripheral blood stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy and filgrastim followed by peripheral stem cell transplantation in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess clinical outcomes, survival, and morbidity of transplantation therapy in patients with chronic myelogenous leukemia when treated with high dose chemotherapy and filgrastim (G-CSF) followed by autologous retrovirally transduced peripheral blood stem cell (PBSC) transplantation.
* Determine whether this priming treatment can increase the fraction of benign Philadelphia chromosome (Ph) negative hematopoietic progenitors in PBSC and reduce the incidence of persistent or recurrent leukemia after autologous transplantation with mobilized PBSC in these patients.
* Assess whether retroviral transduction of mobilized PBSC progenitors determines the contribution of malignant Ph positive progenitors contaminating the graft to relapse after transplantation in these patients.
* Determine whether this priming treatment can expand the benign progenitor population in the PBSC collections from these patients.

OUTLINE: In the priming phase, patients receive cyclophosphamide IV over 2 hours on day 1 and filgrastim (G-CSF) subcutaneously (SQ) daily beginning on day 4 and continuing until the completion of leukapheresis. Peripheral blood stem cells (PBSC) are harvested 4-7 times between days 10 and 21 beginning when blood counts recover (CD34+ cells are selected from 2 of these PBSC collections and transduced with the LN NEO virus prior to cryopreservation).

In the transplant phase, patients who have not received prior radiotherapy receive cyclophosphamide IV over 2 hours daily on days -7 and -6 and total body irradiation on days -4 through -1. Autologous PBSC and LN NEO transduced CD34+ cells are reinfused on day 0. Patients also receive G-CSF IV daily beginning on day 0 and continuing until blood counts recover.

Patients who have received prior radiotherapy receive oral busulfan every 6 hours on days -10 through -7 and cyclophosphamide IV daily on days -6 through -3. Autologous PBSC and LN NEO transduced CD34+ cells are reinfused on day 0. Patients also receive G-CSF IV daily beginning on day 0 and continuing until blood counts recover.

All patients then receive interferon alfa SQ daily until disease progression or unacceptable toxicity.

Patients are followed at 3 weeks; at 3, 6, 9, 12, 18, and 24 months; and then annually thereafter.

PROJECTED ACCRUAL: A total of 4-26 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed chronic or accelerated phase chronic myelogenous leukemia

  * Philadelphia chromosome positive OR
  * BCR/ABL rearrangement
* No blast crisis or post blast crisis
* No moderate to severe fibrosis defined by bilateral trephine biopsies
* Not eligible for or refused to participate in allogeneic marrow transplant protocols
* No splenomegaly (below umbilicus) that does not respond to chemotherapy and/or radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* Karnofsky 90-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Normal organ function (except bone marrow)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior interferon alfa allowed

Chemotherapy:

* Prior hydroxyurea allowed
* At least 2 months since prior busulfan (at time of PBSC harvest)

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M. Verfaillie, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States